CLINICAL TRIAL: NCT05093439
Title: Heart Rate Variabitlity At the Emergency Department: a New Triage Parameter?
Brief Title: Heart Rate Variability At the Emergency Department
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-08267; B.U.N.: B6702020000599 (Other: UZ Gent Ethics Comittee)
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Heart Rate Variability; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients presenting at Emergency Department with severe disease: Participants will be patients with (possible) sepsis, myocardial infarction, cerebrovascular accident, polytrauma or Covid 19 pneumonia who were triaged red or orange following the Manchester triage system.
  Interventions: Diagnostic Test: Heart Rate Variability

INTERVENTIONS:
Diagnostic Test: Heart Rate Variability — Heart rate variability wil be calculated from patients' 10 sec ECG with a dedicated software (Kubios).

SUMMARY:
In this study investigators want to examine if heart rate variability at hospital entry predicts prognosis in participants with severe disease.

DETAILED DESCRIPTION:
Predictive parameters that can predict the outcome are very scarce. Vital parameters such as heart rate, blood pressure, saturation, etc. can be normal for a long time or only slightly changed, even in seriously ill patients. Heart rate variability is a parameter that can be used as a measure of autonomic dysfunction. Lower heart rate variability is associated with increased mortality and morbidity according to recent studies. Heart rate variability could thus be used to identify the need for intervention and treatment more quickly.

In this study, we want to investigate whether there is indeed a relationship between heart rate variability at admission to the emergency department and eventual mortality and morbidity in critically ill patients.

Therefore, heart rate variability will be determined in patients admitted to the emergency department who were triaged in red or orange according to the Manchester Triage System (internationally validated triage system that is also used in the emergency department at UZ Gent). Subanalyses will be made for patients with trauma, sepsis, pneumonia, CVA and acute myocardial infarction. Determination of heart rate variability will be done by EKG monitoring during the first 5 minutes and after 3 hours. There are several parameters that can reflect heart rate variability. Both frequency domain measurements and non-linair measurements will be determined. Use will be made of the Kubios programme, a free programme that can determine these different parameters on the basis of EKG monitoring. Patients who are resuscitated on arrival will be excluded, as well as patients in VKF, as the heart rate variability on arrival cannot be determined for these two groups. Demographic data (age, sex,...), history and home medication, vital parameters (heart rate, blood pressure, saturation, temperature, respiratory rate) and some lab data (lactate, CRP) will also be collected. The primary outcome will be mortality after 30 days. Secondary outcomes that will be studied are the total duration of hospital stay and the duration of stay in the intensive care unit, as well as the need for life-saving interventions (need for surgery, ventilation, inotropics, PCI or thrombolysis).

By collecting these data, we want to find out whether heart rate variability is a good predictor of outcome, and thus the need for ICU admission, faster invasive interventions,... During this study, the patient's management will remain unchanged.

ELIGIBILITY:
Inclusion Criteria:

Patients with (possible) sepsis, myocardial infarction, cerebrovascular accident, polytrauma or Covid 19 pneumonia who were triaged red or orange following the Manchester triage system

Exclusion Criteria:

Patients with cardiac arrest or arrhythmia at arrival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at the Emergency Department with severe disease
Sampling Method: Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days

SECONDARY OUTCOMES:
Length of Hospital Stay | 0 - 100 days
Length of stay at the intensive care unit | 0 - 100 days
Need for life threatening interventions | In 0 - 7 days after admission
  Need for surgery, mechanical ventilation, inotropic medications, PCI or thrombolysis

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent - Emergency Department, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No